CLINICAL TRIAL: NCT03121014
Title: A Phase II Study of Intensity Modulated Total Marrow Irradiation (IM-TMI) in Addition to Fludarabine/Busulfan Conditioning for Allogeneic Transplantation in High Risk AML and Myelodysplastic Syndromes
Brief Title: Study of Intensity Modulated Total Marrow Irradiation (IM-TMI) in Addition to Fludarabine/Busulfan Conditioning for Allogeneic Transplantation in High Risk AML and Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, Hematology, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; fludarabine phosphate; Busulfan; thymoglobulin; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Treatment (Experimental): Patients will receive fludarabine 40 mg/m2 IVBP daily for day -5 (5 days before stem cell infusion) through Day -2, IV busulfan targeting a 4800μM/min/ day from day -5 through day -2, and ATG (Thymoglobulin®) at 0.5 mg/kg IV on day -3, and 2 mg/kg on days -2 and day -1 (Only for recipients of stem cells from unrelated or mismatched donors). In addition to the above conditioning regimen all patients will receive TMI at a dose of 3Gy on days -3, -2 and -1. On day 0, the stem cell product will be infused according to BMT unit policy. Graft versus host disease (GVHD) prophylaxis will consist of administration of tacrolimus and methotrexate. Post-transplant evaluation will be done as per standard care with study data collected at day 30, 60, 90, 180, 365 and 2 years.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: ATG; Radiation: Total Marrow Irradiation; Procedure: Stem Cell Product Infusion; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Fludarabine — 40 mg/m^2 IVBP daily for day -5 (5 days before stem cell infusion) through Day -2
  Other Names: Fludara®
Drug: Busulfan — targeting a 4800μM/min/ day from day -5 through day -2
  Other Names: Busulfex®
Drug: ATG — 0.5 mg/kg IV on day -3, and 2 mg/kg on days -2 and day -1
  Other Names: Thymoglobulin®
Radiation: Total Marrow Irradiation — dose of 3Gy on days -3, -2 and -1
Procedure: Stem Cell Product Infusion — Day 0 according to BMT unit policy
Drug: Tacrolimus — The starting dose is at 0.03 mg/kg/day IV continuous infusion over 24 hr from 4 PM on day -2. Dose will be adjusted to target trough levels of 5-15 ng/mL. More information is available in the protocol document.
  Other Names: FK-506, Prograf®
Drug: Methotrexate — 5mg/m^2 on Day 1, 5 mg/m^2 on Days 3, 6 and 11
  Other Names: Trexall®

SUMMARY:
The study is a Phase II clinical trial. Patients will receive intensity modulated total marrow irradiation (TMI) at a dose of 9 Gy with standard myeloablative fludarabine/ i.v. targeted busulfan (FluBu) conditioning prior to allogeneic hematopoietic stem cell transplant (HSCT).

DETAILED DESCRIPTION:
Patients will receive the following conditioning regimen: fludarabine 40 mg/m2 IVBP daily for day -5 (5 days before stem cell infusion) through Day -2, IV busulfan targeting a 4800μM/min/ day from day -5 through day -2, and ATG (Thymoglobulin®) at 0.5 mg/kg IV on day -3, and 2 mg/kg on days -2 and day -1 (Only for recipients of stem cells from unrelated or mismatched donors). In addition to the above conditioning regimen all patients will receive TMI at a dose of 3Gy on days -3, -2 and -1. On day 0, the stem cell product will be infused according to BMT unit policy. Graft versus host disease (GVHD) prophylaxis will consist of administration of tacrolimus and methotrexate (see Section 8). Post-transplant evaluation will be done as per standard care with study data collected at day 30, 60, 90, 180, 365 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Patients with AML or MDS who meet the following criteria:

   a. Relapsed or refractory AML (including AML in CR2)

   b. Poor-risk AML in first remission, with remission defined as <5% bone marrow blasts morphologically:
   * AML arising from MDS or a myeloproliferative disorder, or secondary AML
   * Poor risk molecular features including presence of FLT3 internal tandem duplication mutation.
   * Poor-risk cytogenetics: Monosomal karyotype, complex karyotype (> 3 abnormalities), inv(3), t(3;3), t(6;9), MLL rearrangement with the exception of t(9;11), or abnormalities of chromosome 5 or 7

     c. Primary refractory disease

     d. MDS with at least one of the following poor-risk features:
   * Poor-risk cytogenetics including 3q abnormalities, 7/7q minus or complex cytogenetics (>3 abnormalities)
   * Current or previous INT-2 or high IPSS score
   * Treatment-related MDS
   * MDS diagnosed before age 21 years
   * Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy
   * Life-threatening cytopenias, including those requiring regular PRBC or platelet transfusions e. CML with a history of accelerated or blast phase
3. Patients must have a related or unrelated peripheral blood stem cell donor as follows:

   1. Sibling donor must be a 6/6 match for HLA-A, -B at intermediate (or higher) resolution and -DRB1 at high resolution using DNA based typing
   2. Unrelated donors must be at least 7/8 match at HLA-A, -B, -C and DRB1 at high resolution using DNA-based typing

Exclusion criteria:

1. Presence of significant co morbidity as shown by:

   1. Left ventricular ejection fraction < 50%
   2. Creatinine clearance <30ml/min
   3. Bilirubin > 2.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST > 5 x ULN
   4. FEV1 and FVC < 50% of predicted or DLCO <50% of predicted once corrected for anemia

   f. Karnofsky score <70 (appendix C)

   g. Hematopoietic cell transplantation comorbidity index >3

   h. Active viral hepatitis or HIV infection

   j. Cirrhosis
2. Pregnancy
3. Patients unable to sign informed consent
4. Patient who have previously received radiation to >20% of bone marrow containing areas.

4. DONOR ELIGIBILITY AND SELECTION

4.1. Donor Selection

Donor evaluation and selection is by standard for normal clinical practice. No study procedures are to be performed on donors. All donors must be willing to donate peripheral blood stem cells and meet institutional or NMDP criteria for donation.

The following prioritization will be used when selecting donors:

1. When possible, an HLA compatible sibling will be used as a donor.
2. For patients who do not have an HLA compatible sibling, an unrelated donor will be used
3. 8/8 matched unrelated donors are preferred over single antigen mismatched donors.

If more than one potential volunteer unrelated donor is considered suitable further selection of the most suitable donor is at the discretion of the treating physician. The following serves only as a guide for prioritization:

1. Age of donor (18-24 > 25-34 > 35-44 > 45+)
2. Sex and parity of donor (male > female, nulliparous female > parous, multiparous female)
3. Cytomegalovirus (CMV) status, if recipient is CMV seronegative (CMV- > CMV+)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival of approximately 30% in high-risk patients conditioned with the Fludarabine/ Busulfan regimen | Up to 1 year
  Using a Simon 2 stage optimal design with α of 0.05 and power of 0.8, 15 patients will be enrolled in the first stage. If greater than 5 patients survive to 1 year without relapse the study will continue into stage 2. Recruitment will then continue to a total of 46 patients. In this expanded cohort, if a total of 18 or more patients survive to 1 year without relapse, the treatment will be judged efficacious and worthy of further study.

SECONDARY OUTCOMES:
Relapse free survival | Up to 1 year
  It will be estimated and reported with 90% confidence intervals. The proportion of patients who are alive at 1-year will also be estimated with a 90% exact binomial confidence interval.
Overall survival | Up to 1 year
  It will be estimated and reported with 90% confidence intervals. The proportion of patients who are alive at 1-year will also be estimated with a 90% exact binomial confidence interval.
Transplant related mortality rate | Up to 1 year
  After accrual of 10 patients, analysis will be performed to ensure that the mortality rate does not exceed 30%. By calculation of confidence intervals to ensure the TRM not exceed 30%, accrual would be halted if n= 6 of 10 (lower bound of the exact, one-sided 90% CI is 35.4%).

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Maahs L, Avila AM, Koshy M, Sweiss K, Ahn KH, Chen Z, Uzoka C, Galvez C, Sanchez M, Rubinstein P, Quigley J, Zucchetti E, Mahmud N, Aydogan B, Patel P, Rondelli D. Intensified conditioning with high-dose total marrow irradiation and myeloablative chemotherapy reduces risk of relapse without increasing toxicity in allogeneic hematopoietic stem cell transplant for high-risk myeloid malignancies: a phase II study. Haematologica. 2026 Jan 1;111(1):177-183. doi: 10.3324/haematol.2025.287457. Epub 2025 Jun 19. PMID 40534485